CLINICAL TRIAL: NCT03029585
Title: Phase II Study of Four Dose Levels of Intraperitoneal NanoPac® Plus IV Carboplatin and Paclitaxel in Patients With Epithelial Ovarian Cancer Undergoing Cytoreductive Surgery
Brief Title: Phase II Study of Intraperitoneal NanoPac® in Patients With Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: NanOlogy, LLC (Industry)
Collaborators: US Biotest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NANOPAC-2016-01
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: Ovarian Carcinoma
Keywords: ovarian carcinoma; ovarian cancer; ovarian neoplasms; ovarian diseases
MeSH Terms: conditions — Ovarian Neoplasms; Ovarian Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- NanoPac® 100 mg/m2 (Experimental): Intraperitoneal NanoPac® 100 mg/m2 applied immediately post-cytoreductive surgery, followed by standard of care intravenous chemotherapy.
  Interventions: Drug: NanoPac® 100 mg/m2; Drug: Standard of Care Intravenous Chemotherapy
- NanoPac® 200 mg/m2 (Experimental): Intraperitoneal NanoPac® 200 mg/m2 applied immediately post-cytoreductive surgery, followed by standard of care intravenous chemotherapy.
  Interventions: Drug: NanoPac® 200 mg/m2; Drug: Standard of Care Intravenous Chemotherapy
- NanoPac® 300 mg/m2 (Experimental): Intraperitoneal NanoPac® 300 mg/m2 applied immediately post-cytoreductive surgery, followed by standard of care intravenous chemotherapy.
  Interventions: Drug: NanoPac® 300 mg/m2; Drug: Standard of Care Intravenous Chemotherapy
- NanoPac® 400 mg/m2 (Experimental): Intraperitoneal NanoPac® 400 mg/m2 applied immediately post-cytoreductive surgery, followed by standard of care intravenous chemotherapy.
  Interventions: Drug: NanoPac® 400 mg/m2; Drug: Standard of Care Intravenous Chemotherapy
- Standard of Care Intravenous Chemotherapy (Active Comparator): Standard of care intravenous chemotherapy (with platinum and taxane agents) administered per institutional standards.
  Interventions: Drug: Standard of Care Intravenous Chemotherapy

INTERVENTIONS:
Drug: NanoPac® 100 mg/m2 — Single intraperitoneal injection of 100 mg/m2 NanoPac® during cytoreductive surgery, followed by standard-of-care IV carboplatin and IV paclitaxel treatment
  Arms: NanoPac® 100 mg/m2
Drug: NanoPac® 200 mg/m2 — Single intraperitoneal injection of 200 mg/m2 NanoPac® during cytoreductive surgery, followed by standard-of-care IV carboplatin and IV paclitaxel treatment
  Arms: NanoPac® 200 mg/m2
Drug: NanoPac® 300 mg/m2 — Single intraperitoneal injection of 300 mg/m2 NanoPac® during cytoreductive surgery, followed by standard-of-care IV carboplatin and IV paclitaxel treatment
  Arms: NanoPac® 300 mg/m2
Drug: NanoPac® 400 mg/m2 — Single intraperitoneal injection of 400 mg/m2 NanoPac® during cytoreductive surgery, followed by standard-of-care IV carboplatin and IV paclitaxel treatment
  Arms: NanoPac® 400 mg/m2
Drug: Standard of Care Intravenous Chemotherapy — Cytoreductive surgery followed by standard-of-care IV carboplatin and IV paclitaxel treatment

SUMMARY:
This study will evaluate NanoPac® administered intraperitoneally (IP) immediately post-cytoreductive surgery, followed by standard of care (SOC) intravenous (IV) chemotherapy, in women with ovarian cancer. The study will compare IP NanoPac® (plus IV chemotherapy) with SOC IV chemotherapy alone.

DETAILED DESCRIPTION:
Research has shown that the administration of chemotherapy directly into the peritoneal cavity (intraperitoneal [IP] chemotherapy) may provide a significant survival benefit to women with ovarian cancer when combined with cytoreductive surgery and IV chemotherapy.

This study will include a dose-finding phase and an efficacy phase to evaluate IP NanoPac® administered immediately post-cytoreductive surgery in women with ovarian cancer. In the dose-finding phase, subjects will be enrolled in dose-escalated cohorts of three subjects and receive IP NanoPac® at 100, 200, 300, or 400 mg/m2 plus standard of care (SOC) IV chemotherapy. Subjects will be followed for disease status for 12 months. The two best doses from the dose-finding phase will be determined. In the efficacy phase, subjects will be randomized 1:1:1 to one of the two best doses plus SOC IV chemotherapy or SOC alone.

ELIGIBILITY:
Inclusion Criteria:

* Epithelial ovarian cancer which is contained within the abdomen, but may include pleural effusion if that is the limit of non-peritoneal cavity disease. If subject has recurrent epithelial ovarian cancer, the disease must be platinum sensitive (recurrence >6 months from prior chemotherapy regimen that included a platinum agent and cytoreductive surgery)
* Subject appropriate for cytoreductive surgery and treatment with IV platinum and paclitaxel
* Minimal or non-symptomatic ascites
* ≥18 years old
* Signed informed consent

Exclusion Criteria:

* Epithelial ovarian cancer outside of the peritoneal cavity, with the exception of pleural effusions
* Anticipated use of concomitant chemotherapy (other than the protocol-specified agents), immunotherapy, or radiation therapy
* Treatment with a prior investigational agent within 30 days of planned instillation of NanoPac®, with the exception of subjects participating in poly (ADP-ribose) polymerase (PARP) inhibitor trials. These subjects must discontinue the investigational agent prior to surgery
* Known sensitivity to any of the study medication components or the chemotherapy regimen
* History of prior malignancy other than ovarian that has not been in remission for >5 years, with the exception of basal cell or squamous cell carcinoma or cervical carcinoma in situ on biopsy
* Ileostomy or hepatic resection during current cytoreductive surgery
* Women of childbearing potential not practicing adequate forms of birth control

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Walker, MD, Principal Investigator — University of Oklahoma; Gere diZerega, MD, Study Chair — US Biotest, Inc./NanOlogy, LLC
Locations (7):
- United States (7):
  - University of Chicago, Chicago, Illinois
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - SUNY Downstate, Brooklyn, New York
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NanoPac® 100 mg/m2 | NanoPac® 200 mg/m2
Started | 7 | 3
Completed | 5 | 2
Not Completed | 2 | 1
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NanoPac® 100 mg/m2 | NanoPac® 200 mg/m2 | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Continuous [Median (Full Range); unit: years] | 68 [50 to 72] | 62 [56 to 71] | 67 [50 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Disease Status [Count of Participants; unit: Participants]
  Primary | 4 | 2 | 6
  Recurrent | 3 | 1 | 4
ECOG Status [Count of Participants; unit: Participants] — ECOG Performance Scale:
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    ECOG 0 | 5 | 2 | 7
    ECOG 1 | 2 | 1 | 3
Status of Ovarian Cancer at Screening [Count of Participants; unit: Participants] — Ovarian cancer stages range from stage I (1) through IV (4). As a rule, the lower the number, the less the cancer has spread. A higher number, such as stage IV, means cancer has spread more.
  Participants
    IIIA2 | 0 | 1 | 1
    IIIB | 2 | 0 | 2
    IIIC | 4 | 1 | 5
    IVB | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events
Description: Adverse events will include any clinically relevant changes in laboratory values, vital signs, and physical examination. Treatment-emergent adverse events occur when the date and time of the adverse event onset is on or after the first application of the investigational agent and any time up to when the intravenous chemotherapy commences. Treatment-emergent adverse events will be summarized for each treatment group. The summaries will include an overall summary of the number of subjects reporting and the number of events reported, summaries of adverse events leading to termination or death, and summaries by severity and relatedness (separately and combined). Of greatest interest will be post-surgery signs of toxicity (e.g., severe abdominal pain after 5-7 days, neutropenia, thrombocytopenia, bowel dehiscence, prolonged ileus).
Time Frame: 12 months
Measure: Number; unit: Treatment Emergent Adverse Events
Arm/Group | NanoPac® 100 mg/m2 | NanoPac® 200 mg/m2
Number analyzed (Participants) | 7 | 3
Treatment Emergent Adverse Events | 80 | 28

2. Secondary Outcome: Maximum Plasma Concentration of Paclitaxel (Cmax)
Description: Plasma samples will be taken on Day 1 at 1, 2, 4, 8, and 24 hours post-intraperitoneal administration of NanoPac® and weekly thereafter until IV chemotherapy begins. Additionally, a pharmacokinetics (PK) sample will be collected from every subject prior to each cycle of IV chemotherapy for determination of paclitaxel concentrations to assess potential NanoPac® persistence. PK levels of paclitaxel in the plasma will be summarized descriptively.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | NanoPac® 100 mg/m2 | NanoPac® 200 mg/m2
Number analyzed (Participants) | 7 | 3
ng/mL | 12.56 (10.98) | 26.50 (13.56)

3. Secondary Outcome: Progression Free Survival (PFS) at 12 Months
Description: Progression free survival (PFS) was assessed every 3 months until the end of the 12-month follow-up period, and every 6 months thereafter until progression or the last subject in the trial has completed 12 months of follow-up. Factors taken into account to determine time-to-progression included CA-125 levels, tumor burden as assessed by imaging and utilizing RECIST version 1.1 for assessment of response, and cancer-related symptoms such as bowel obstruction and ascites.
Time Frame: 12 months post-treatment
Population: Of the 10 subjects enrolled, four subjects were not evaluable for PFS at 12 months post-NanoPac instillation. For one subject, no imaging was performed over the course of the study; one subject was deceased due to leptomeningeal carcinomatosis; one subject was deceased due to a respiratory arrest; and one subject withdrew consent from the study. Both deaths were considered not related to study medication by the Investigator and the Medical Monitor.
Measure: Count of Participants; unit: Participants
Arm/Group | NanoPac® 100 mg/m2 | NanoPac® 200 mg/m2
Number analyzed (Participants) | 4 | 2
Participants
  PFS at 12 months | 4 | 0
  Disease Progression | 0 | 2

ADVERSE EVENTS:
Time Frame: AEs were collected at all study visits from the time of dosing until end of study, for a planned 30-month collection period for each subject.
Arm/Group | NanoPac® 100 mg/m2 | NanoPac® 200 mg/m2
All-Cause Mortality (participants affected / at risk) | 1/7 | 1/3
Serious Adverse Events (participants affected / at risk) | 4/7 | 3/3
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NanoPac® 100 mg/m2 (N=7) | NanoPac® 200 mg/m2 (N=3)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pelvic fluid collection (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NanoPac® 100 mg/m2 (N=7) | NanoPac® 200 mg/m2 (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (5) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (5) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (2)
Administration site extravasation (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (5) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0)
Blood chloride decreased (Investigations) | 1 (1) | 0 (0)
Blood urea decreased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 1 (1) | 0 (0)
Lymphocyte count (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Protein total decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count increased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Hypokalacaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic fluid collection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT03029585/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/85/NCT03029585/SAP_001.pdf